CLINICAL TRIAL: NCT01494909
Title: Development Of An Innovative Panel of Methods To Measure Intestinal Macronutrient Digestion, Absorption, and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Arkansas Children's Hospital Research Institute (Other); University of Arkansas (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 113047
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis
Keywords: protein digestion; fat absorption; gut function; glucose absorption; CF; pancreatic intake; feeding
MeSH Terms: conditions — Cystic Fibrosis | interventions — Ensure Plus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ensure plus (Experimental): Ensure sip feeds during 6 hours. After 2 hours pancreatic intake
  Interventions: Dietary Supplement: Ensure plus

INTERVENTIONS:
Dietary Supplement: Ensure plus — Ensure plus sip feeds every 20 min during 6 hours. After 2 hour pancreatic enzyme intake in CF

SUMMARY:
Malnutrition is a significant problem in children and adults with Cystic fibrosis (CF). An impaired intestinal digestion and absorption capacity is one of the main factors responsible for the malnutrition in CF. This impairment starts early in life, leading to malnutrition, muscle weakness, impaired immune and lung function associated with poor prognosis. As low BMI and body weight is strongly associated with morbidity and mortality, a reduction in weight loss in CF and its manifestations would save the healthcare system substantially per year. Simple methods to measure the digested portions and utilization of nutrients and the effectiveness of pancreatic enzyme preparations and medications in CF are not available. Developing a panel of methods to accurately measure gut digestion, absorption and function will lead to studies optimizing nutritional regimen and pancreatic enzyme replacement therapy in CF. Furthermore, it will provide detailed insight in the disease and age related mechanisms of gut dysfunction in CF. Finally, it will provide required information that will lead to implement new strategies to improve gut health in order to enhance nutritional status, quality of life and survival.

The hypothesis is that intestinal macronutrient digestion, absorption and function in CF can be quantified by an innovative panel of methods using stable isotopes. With this panel of methods, information can be obtained on the effect of disease progression on lipid, protein and glucose digestion and absorption and on gut function in CF as well as in other diseases and conditions characterized by a compromised gut. Furthermore, the optimal nutritional regimen and pancreatic enzyme therapy if applicable can be evaluated in these diseases. In the present study the investigators will study: 1. Pediatric patients with CF at Arkansas Children's Hospital; 2. Adult patients with CF at University of Arkansas for Medical Sciences. 3. Healthy control subjects. Diagnosis of CF is made based on universal diagnostic criteria. All CF patients are characterized by abnormal lipid digestion based on clinical and or laboratory (72 hour fat analysis or fecal elastase measurement) diagnosis, and requiring pancreatic enzyme replacement therapy, and no presence of unstable metabolic diseases. Additional criteria for the CF pediatric inpatients are: admitted to ACH for treatment of exacerbations of CF disease, clinically stable. The CF outpatients are stable outpatients with pancreatic insufficiency.

ELIGIBILITY:
Inclusion Criteria:

Adult subjects with CF

1. Diagnosis of CF based on universal diagnostic criteria
2. Pancreatic insufficiency based on clinical diagnosis
3. Abnormal lipid digestion requiring pancreatic enzyme replacement therapy
4. Age is 18 years and older.
5. Admitted to UAMS for treatment of exacerbations of CF (inpatients) or under routine medical control at the CF center of UAMS
6. Clinically stable CF at the time of enrollment

Healthy adults

1. Age is 18 years and older at the time of enrollment.
2. BMI between 18 and 35 kg/m2

Exclusion Criteria:

Pediatric and adult CF groups

1. Unstable metabolic diseases including liver (cirrhosis) or renal disease
2. Chronic respiratory failure with cor pulmonale
3. Any other condition according to the principle investigator or study physician would interfere with proper conduct of study / safety of the patient
4. Failure to give assent / informed consent
5. Diagnosis of severe lung disease, defined as FEV1 < 35% predicted

Healthy adults

* Presence of acute or chronic unstable diseases such as liver, renal, heart or lung disease
* Previous surgery less than 4 weeks prior to the experiment
* Recent involuntary weight loss (>10% in the past 3 months)
* Any documented autoimmune disease
* Any other condition according to the principle investigator or study physician would interfere with collecting study samples
* Failure to give informed consent

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-11-15 (Actual); Primary Completion 2011-12-07 (Actual); Study Completion 2011-12-07 (Actual)

PRIMARY OUTCOMES:
Fatty acid absorption during feeding and effect pancreatic enzyme intake | 8 hours
  Enrichment in palmitic acid and tripalmitin fatty acids in plasma

SECONDARY OUTCOMES:
Protein digestion during feeding and effect pancreatic enzyme intake | 8 hours
  Ratio enrichment in plasma free phenylalanine vs from protein spirulina
Glucose absorption during feeding and effect pancreatic enzyme intake | 8 hours
  Plasma and urine 3-O-methyl-D-glucose

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas EP Deutz, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Engelen MP, Com G, Anderson PJ, Deutz NE. New stable isotope method to measure protein digestibility and response to pancreatic enzyme intake in cystic fibrosis. Clin Nutr. 2014 Dec;33(6):1024-32. doi: 10.1016/j.clnu.2013.11.004. Epub 2013 Nov 9. PMID 24268783